CLINICAL TRIAL: NCT02944110
Title: Delineation of the Diabetogenic Role of Extrapancreatic Glucagon in Totally Pancreatectomised Patients Using Glucagon Receptor Antagonism
Acronym: PX-GRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15009763
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Diabetes After Total Pancreatectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pancreatectomised + LY2409021 (Active Comparator): During the experimental day the patient will undergo a 75gr-OGTT. On the evening before the experimental day, the patient will ingest a dose of 300mg of LY2409021.
  Interventions: Drug: Glucagon receptor antagonist LY2409021
- Pancreatectomised + placebo (Placebo Comparator): During the experimental day the patient will undergo a 75gr-OGTT. On the evening before the experimental day, the patient will ingest placebo tablets.
  Interventions: Drug: Placebo
- Healthy + LLY2409021 (Active Comparator): During the experimental day the subject will undergo a 75gr-OGTT. On the evening before the experimental day, the subject will ingest a dose of 300mg of LY2409021.
  Interventions: Drug: Glucagon receptor antagonist LY2409021
- Healthy + placebo (Placebo Comparator): During the experimental day the subject will undergo a 75gr-OGTT. On the evening before the experimental day, the subject will ingest placebo tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucagon receptor antagonist LY2409021 — single oral dose of 300mg
  Arms: Healthy + LLY2409021; Pancreatectomised + LY2409021
Drug: Placebo — Oral dose of placebo tablets
  Arms: Healthy + placebo; Pancreatectomised + placebo

SUMMARY:
Patients with diabetes are characterised not only by compromised insulin secretion and action, but also by elevated plasma levels of the 29-amino acid peptide hormone glucagon, which hitherto has been considered a pancreas-derived hormone (produced in and secreted from alpha cells in the islets of Langerhans). In patients with diabetes, circulating glucagon concentrations are elevated in the fasting state and fail to decrease appropriately or even increase in response to an oral glucose tolerance test (OGTT) or after ingestion of a mixed meal. Hyperglucagonaemia is known to be a potent stimulator of hepatic glucose output, and, thus, contributes significantly to the fasting and postprandial hyperglycaemia characterising patients with diabetes. Despite intense research over the years the mechanisms behind the elevated glucagon levels in diabetes is still not clear. Recently, the investigators showed that totally pancreatectomised patients also show a hyperglucagonaemic response during OGTT, a finding that suggests that the pancreas is not the only source of glucagon production in man.

In the present project, the investigators wish to evaluate the impact of gastrointestinally derived glucagon secretion observed in totally pancreatectomised patients on postprandial glucose tolerance.

The investigators hypothesise that antagonisation of glucagon signalling (from gastrointestinally derived glucagon) in totally pancreatectomised patients will improve or perhaps normalise the patients glucose tolerance during a 75g-OGTT. In order to test this hypothesis, the investigators wish to apply the potent and selective oral antagonist of the human glucagon receptor LY2409021 and placebo, respectively.

The study is a randomised, placebo-controlled, double-blinded, cross-over study.

10 healthy persons and 10 pancreatectomized patients (i.e. patients who have had their pancreata removed due to pancreatic cancer or severe chronic pancreatitis) will be subjected to two experimental days with LY2409021 and placebo, respectively, on which they will undergo an OGTT followed by a fasting period and finished off with an ad libitum meal.

ELIGIBILITY:
Inclusion criteria

Pancreatectomised patients

* Caucasian above 18 years of age who have undergone total pancreatectomy
* Normal haemoglobin
* Informed consent

Healthy subjects

* Normal fasting plasma glucose and normal HbA1C (according to the World Health Organization (WHO) criteria)
* Normal haemoglobin
* Age above 18 years
* Informed consent

Exclusion criteria

Pancreatectomised patients

* Inflammatory bowel disease
* Operation within the last 3 months
* Ongoing chemotherapy or chemotherapy within the last 3 months
* Gastrointestinal resection (other than the gastro-duodenectomy performed in connection with total pancreatectomy) and/or ostomy
* Nephropathy (serum creatinine >150 µmol/l and/or albuminuria)
* Severe liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >3× normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years
* Uncontrolled hypertension and/or significant cardiovascular disease
* Any condition that the investigator feels would interfere with trial participation

Healthy subjects

* Diabetes or prediabetes (according to the WHO criteria)
* First-degree relatives with diabetes
* Inflammatory bowel disease
* Gastrointestinal resection and/or ostomy
* Nephropathy (serum creatinine >150 µM and/or albuminuria
* Liver disease (ALAT and/or serum ASAT >2×normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
PPG excursions measured as incremental area under curve (iAUC) | -120,-45,-30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes

SECONDARY OUTCOMES:
differences in gastric emptying, measurement of s-paracetamol | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
  measurement of time to peak and incremental area under the curve (iAUC)
food intake and appetite | at time 0,30,60,90,120,150,180 minutes
  assessed by a visual analogue scale
resting energy expenditure (REE) | -90,30,150 minutes
  measured by calorimetry
p-glucose mmol/L | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
glucagon pmol/l | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
free fatty acids μmol/l | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
p-triglyceride mmol/l | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
Amino Acid concentration μmol/l | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
  total and fractionated
cholecystokinin pmol/l | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes
Gastric inhibitory peptide (GIP) and Glucagon like peptide-1 (GLP-1) pmol/l | -30,-15,0,5,10,15,20,25,30,40,50,60,70,80,90,105,120,135,150,180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, Professor, Principal Investigator — Head of department at Center for Diabetes Research, Gentofte Hospital, Kildegaardsvej 28, 2900 Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juel CT, Lund AB, Haedersdal S, Andersen MM, Hansen CP, Storkholm JH, van Hall G, Hartmann B, Rosenkilde MM, Kibsgaard CJ, Dela F, Albrechtsen NJW, Holst JJ, Vilsboll T, Knop FK. Using glucagon receptor antagonism to evaluate the physiological effects of extrapancreatic glucagon in totally pancreatectomised individuals: a randomised controlled trial. Diabetologia. 2025 Dec;68(12):2807-2822. doi: 10.1007/s00125-025-06534-z. Epub 2025 Sep 18. PMID 40968190
- [Derived] Juel CTB, Dejgaard TF, Hansen CP, Storkholm JH, Vilsboll T, Lund A, Knop FK. Glycemic Control and Variability of Diabetes Secondary to Total Pancreatectomy Assessed by Continuous Glucose Monitoring. J Clin Endocrinol Metab. 2021 Jan 1;106(1):168-173. doi: 10.1210/clinem/dgaa731. PMID 33053154